## **English Version**

| Dear |
|------|

We invite you to the study titled "The effect of auricular vagus nerve stimulation on pain and quality of life in patients with Fibromyalgia Syndrome" directed by Nazlı Kutlu, Bahçeşehir University graduate student. Before deciding whether or not to participate in this research, you need to know why the research was done, the benefits and risks it will bring to you. For this reason, it is important to read and understand this form. Read the information below carefully and ask the researcher if there are places you do not understand or want more information.

Participating in the research is completely voluntary. You have the right not to participate in the study or to quit at any time.

Purpose of the research:

The aim of this study is to investigate the effect of exercise applications with auricular vagus nerve stimulation on common pain in people who experience pain related to fibromyalgia at certain intervals but have not received any treatment for this pain.

The method and procedures to be followed:

The aim of the study; To evaluate the effect of auricular vagus nerve stimulation applied to patients with fibromyalgia syndrome (FMS) in addition to exercise therapy on pain and quality of life. For this purpose, 60 female patients between the ages 18-50, who are diagnosed with FMS according to the ACR 2010 diagnostic criteria, will be randomly divided into 2 groups of 30 people. Exercise treatment in the form of 20 sessions home program for the first group, 20 sessions in the form of 20 sessions home program in addition to the exercise treatment in the form of 20 sessions home program. and its frequency is 10 Hz. auricular vagus nerve stimulation will be applied. Patients before and after treatment; Visual Analogue Scale (VAS) for pain, Beck Depression Scale for depression, Beck Anxiety Scale for anxiety, FIQ for functional evaluation, and SF-36 for quality of life.

You are expected to provide clear answers to the questions that will be asked during the evaluation.

| l | (Name-surname | of the volunteer) |
|---|---------------|-------------------|
|---|---------------|-------------------|

I have read all the comments on the Informed Volunteer Consent Form. The written and verbal explanation to me about the research mentioned above and its purpose was made by the researcher mentioned below. I fully accepted the scope and purpose of the work I was asked to participate in, voluntarily my responsibilities. I know that I voluntarily participated in the research, I can leave the research with or without justification at any time, and I can

be excluded from the research by the researcher, regardless of my own will. In these conditions, the said research; I agree to participate with my own consent without any influence.

| The researcher's; |
|------------------------------|
| Name Surname: Nazlı Kutlu |
| Phone Number: 0531 835 14 52 |
| Volunteer's |
| Name and surname: |
| Phone number: |
| Signature: |
| Date: |
| Turkish Version: |
| Sayın |

Sizi Bahçeşehir Üniversitesi Yüksek Lisans öğrencisi Nazlı Kutlu tarafından yönetilen "Fibromiyalji Sendromlu hastalarda auriküler vagus sinir uyarımının ağrı ve yaşam kalitesi üzerine etkisi" başlıklı araştırmaya davet ediyoruz. Bu araştırmaya katılıp katılmama kararını vermeden önce , araştırmanın neden yapıldığını, size getireceği fayda ve riskleri bilmeniz gerekmektedir. Bu nedenle bu formun okunup anlaşılması önemlidir. Aşağıdaki bilgileri dikkatlice okuyunuz anlamadığınız veya daha fazla bilgi almak istediğiniz yerler olursa araştırmacıya sorunuz.

Araştırmaya katılmak tamamen gönüllülük esasına dayanmaktadır. Çalışmaya katılmama veya herhangi bir anda çalışmadan çıkma hakkına sahipsiniz.

## Araştırmanın Amacı:

Bu araştırmanın amacı, günlük yaşamında belirli aralıklarla fibromiyaljiye bağlı ağrı şikayetleri yaşayan fakat bu ağrısına yönelik herhangi bir tedavi görmemiş kişilerde aurikular vagus sinir stimülasyonuyla egzersiz uygulamalarının yaygın ağrılar üzerindeki etkisinin araştırılmasıdır.

İzlenecek olan yöntem ve yapılacak işlemler:

Çalışmanın amacı; Fibromiyalji sendromlu (FMS) hastalarda egzersiz tedavisine ek olarak uygulanan auriküler vagus sinir uyarımının ağrı ve yaşam kalitesine etkisini değerlendirmektir. Bu amaçla, ACR 2010 tanı kriterlerine göre FMS tanısı konan, 18-50 yaş arası, 60 kadın hasta rastgele yöntemle 30'ar kişilik 2 gruba ayrılacaktır. 1. gruba 20 seans ev programı şeklinde egzersiz tedavisi , 2. gruba 20 seans ev programı şeklinde egzersiz

tedavisine ek olarak 20 seans günde 20 dk. ve frekansı 10 Hz. olacak şekilde auriküler vagus sinir stimülasyonu uygulanacaktır. Olgular tedavi öncesi ve sonrası; ağrı açısından Vizüel Analog Skalası (VAS), depresyon açısından Beck Depresyon Ölçeği, anksiyete açısından Beck Anksiyete Ölçeği, fonksiyonel değerlendirme açısından FIQ ve yaşam kalitesi açısından SF-36 ile değerlendirilecektir.

Sizden beklenen değerlendirme sırasında sorulcak olan sorulara açık ve net cevaplar vermenizdir.

| Ben | .( | gör | nüllü | nün | adı- | soya | ıdı) |
|-----|----|-----|-------|-----|------|------|------|
|-----|----|-----|-------|-----|------|------|------|

Bilgilendirilmiş Gönüllü Olur Formundaki tüm açıklamaları okudum. Bana, yukarıda konusu ve amacı belirtilen araştırma ile ilgili yazılı ve sözlü açıklama aşağıda belirtilen araştırmacı tarafından yapıldı. Katılmam istenen çalışmanın kapsamını ve amacını, gönüllü olarak üzerime düşen sorumlulukları tamamen kabul ettim. Araştırmaya gönüllü olarak katıldığımı, istediğim zaman gerekçeli veya gerekçesiz olarak araştırmadan ayrılabileceğimi ve kendi isteğime bakılmaksızın araştırmacı tarafından araştırma dışı bırakılabileceğimi biliyorum. Bu koşullarda söz konusu araştırmaya; baskı ve zorlama olmaksızın kendi rızamla katılmayı kabul ediyorum.

## Araştırmacının;

Adı Soyadı: Nazlı Kutlu

Telefon Numarası: 0531 835 14 52

Gönüllünün;

Adı Soyadı:

Telefon Numarası:

İmzası:

Tarih: